CLINICAL TRIAL: NCT06162832
Title: Evaluation of Clinical and Radiographic Parameters in Bony Defects Treated With Recombinant Human Platelet-derived Growth Factor in Combination With Allograft
Brief Title: Periodontal Regeneration With Recombinant Human Platelet Derived Growth Factor (rH-PDGF-BB) and Allograft
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Collaborators: LifeNet Health (Industry); Lynch Biologics LLC (Industry)
Responsible Party: Principal Investigator, Jesus Israel Rodríguez Pulido, Doctor, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPSI-010613
Record Dates: First submitted 2023-06-22; First posted 2023-12-08 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Periodontal Diseases
Keywords: Periodontal Regeneration; Grow Factors; intraosseous defects
MeSH Terms: conditions — Periodontal Diseases | interventions — Transplantation, Homologous; Becaplermin; Saline Solution

STUDY DESIGN:
Intervention Model Description: The study was conducted in two groups with control and experimental groups which were evaluated during a period of six months with monthly evaluation until the results were obtained.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: It is a triple-blind study, where the operator, the investigator and the statistician have no knowledge of the material placed in the procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Allograft (Active Comparator): Will be used Demineralized cancellous allograft 250-1000um
  Interventions: Combination Product: Allograft and rHPDGF-BB; Combination Product: Allograft and Saline solution
- Saline Solution (Sham Comparator): The saline solution will be used for hydrate the bone graft 20 minutes before the placement at the defect
  Interventions: Combination Product: Allograft and Saline solution
- rhPDGF-BB (GEM21, Lynch Biologics) (Experimental): The rhPDGF-BB will be used for hydrate the bone graft 20 minutes before the placement at the defect
  Interventions: Combination Product: Allograft and rHPDGF-BB

INTERVENTIONS:
Combination Product: Allograft and rHPDGF-BB — At this intervention the periodontal defect will be treated with allograft and rHPDGF-BB (GEM21)
  Other Names: GEM21; Allograft
  Arms: Allograft; rhPDGF-BB (GEM21, Lynch Biologics)
Combination Product: Allograft and Saline solution — This will be used as the control group
  Arms: Allograft; Saline Solution

SUMMARY:
Growth factors are defined as small proteins that trigger a cellular response after binding to cell receptors; Tissue engineering is now clinically applicable in a commercially available system involving the use of recombinant human platelet-derived growth factor.

The objective of this study is to evaluate clinical and radiographic parameters in bone defects treated with platelet-derived growth factor in combination with allograft.

Our hypothesis: Defects treated with DFDBA and rhPDGF-BB have better clinically and radiographic results that the defects treated with DFDBA and saline solution.

DETAILED DESCRIPTION:
The study will be performed in 30 periodontal defects of 2 and 3 walls. The experimental group will consist of DFDBA placement with rhPDGF-BB and control DFDBA with saline solution. The clinical parameters recorded were Probing deep (PD), clinical attachment level (CAL), recession depth, Index of bleeding and plaque at baseline and at six months. Our universe is patients with periodontitis attending at the clinical in Periodontics at the Autonomous University of Nuevo Leon (UANL) School of Dentistry.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of periodontitis
* Infrabony defects of 2 walls, 3 walls and combined defects
* Patients ASA (American Society of Anesthesiologists) I and II
* Patients who smoke less than 10 cigarettes

Exclusion Criteria:

* Patients undergoing bisphosphonate therapy
* Furcation defects
* Patients with evidence of blood dyscrasias.
* Pregnant patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-07-16 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Probing depth | Initial and six months after surgery
  The distance from free gingival margin to sulcus depth, ≥4 millimeters (mm)
Bleeding on probing | Initial and six months after surgery
  Method to asses gingival inflammation. Gingival health is defined as < 10% bleeding sites
Gingival Recession | Initial and six months after surgery
  The distance from the soft tissue (gingiva or alveolar mucosa) margin to cemento-enamel junction, ≥1 millimeters (mm)
Clinical Attachment Level | Initial and six months after surgery
  The distance from the cemento-enamel junction to the tip of a periodontal probe during periodontal diagnostic probing, ≥2 mm (millimeters)
Gingival Phenotype | Initial and six months after surgery
  Gingival phenotype is determined by gingival thickness and keratinized tissue width.
  Probe visible: thin (≤1 mm). Probe not visible: thick (>1mm).
Plaque control record | Initial and six months after surgery
  O'Leary index is used for assessing oral hygiene skills of the patient
Radiographic Measurements | Initial and six months after surgery
  Cemento-enamel junction (CEJ)-Defect Base (DB): The distance of the cementoenamel junction at the base of the defect.
  Cemento-enamel junction (CEJ)-Bone crest (BC): The distance of the cemento-enamel junction to the crest of bone.
  Cemento-enamel junction (CEJ)- Root apex (RA): The distance of the cemento-enamel junction to root apex.
  Lineal Bone Growth (LBG) = CEJ to base of defect at baseline - CEJ to base of defect at 6 months.
  %BF: Percent bone fill was calculated by dividing LBG by the depth of the original bone defect

CONTACTS AND LOCATIONS:
Overall Officials: Jessica P Arredondo Muñoz, Resident, Principal Investigator — Posgrado De Periodoncia, Universidad autónoma de Nuevo León; Maria Fernanda Treviño Campa, Resident, Principal Investigator — Posgrado De Periodoncia, Universidad autónoma de Nuevo León; Gloria Martínez Sandoval, DR, Study Director — Posgrado De Periodoncia, Universidad autónoma de Nuevo León; Norma I Rodríguez Franco, DR, Study Director — Posgrado De Periodoncia, Universidad autónoma de Nuevo León; Jesús I Rodríguez Pulido, DR, Principal Investigator — Posgrado De Periodoncia, Universidad autónoma de Nuevo León; Andrea Ravidà, DDS, MS, Study Chair — Department of Periodontics and Preventive Dentistry, University of Pittsburgh School of Dental Medicine
Locations (1):
- Posgrado de Periodoncia, Facultad de Odontología, Universidad Autónoma de Nuevo León, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McClain PK. The use of recombinant human platelet-derived growth factor-BB in combination with beta-tricalcium phosphate and rhPDGF-BB in combination with freeze-dried bone allograft plus barrier in two separate complex infrabony defects with long-term follow-up. Clin Adv Periodontics. 2022 Dec;12(4):256-261. doi: 10.1002/cap.10212. Epub 2022 Oct 25. PMID 36281628
- [Background] Nevins M, Camelo M, Nevins ML, Schenk RK, Lynch SE. Periodontal regeneration in humans using recombinant human platelet-derived growth factor-BB (rhPDGF-BB) and allogenic bone. J Periodontol. 2003 Sep;74(9):1282-92. doi: 10.1902/jop.2003.74.9.1282. PMID 14584860
- [Result] Nevins M, Giannobile WV, McGuire MK, Kao RT, Mellonig JT, Hinrichs JE, McAllister BS, Murphy KS, McClain PK, Nevins ML, Paquette DW, Han TJ, Reddy MS, Lavin PT, Genco RJ, Lynch SE. Platelet-derived growth factor stimulates bone fill and rate of attachment level gain: results of a large multicenter randomized controlled trial. J Periodontol. 2005 Dec;76(12):2205-15. doi: 10.1902/jop.2005.76.12.2205. PMID 16332231
- [Result] Nevins M, Kao RT, McGuire MK, McClain PK, Hinrichs JE, McAllister BS, Reddy MS, Nevins ML, Genco RJ, Lynch SE, Giannobile WV. Platelet-derived growth factor promotes periodontal regeneration in localized osseous defects: 36-month extension results from a randomized, controlled, double-masked clinical trial. J Periodontol. 2013 Apr;84(4):456-64. doi: 10.1902/jop.2012.120141. Epub 2012 May 21. PMID 22612364